CLINICAL TRIAL: NCT01739478
Title: Packing of Perianal Abscess Cavities (PPAC) Trial: A Randomised Multicentre Trial Comparing Packing With Non-packing of the Abscess Cavity
Brief Title: Packing of Perianal Abscess Cavities Trial: A Randomised Multicentre Trial Comparing Packing With Non-packing of the Abscess Cavity
Acronym: PPAC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: North Western Research Collaborative (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: NWRC-PPAC
Record Dates: First submitted 2012-11-29; First posted 2012-12-03 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-12

CONDITIONS: Perianal Abscess

ARMS (2):
- Non-packing of abscess cavity (Experimental)
  Interventions: Other: External dressing
- Packing of abscess cavity (Other): Current practice
  Interventions: Other: Packing of abscess cavity; Other: External dressing

INTERVENTIONS:
Other: Packing of abscess cavity
  Arms: Packing of abscess cavity
Other: External dressing — Application of external dressing whilst abscess cavity heals

SUMMARY:
The aim of this study is to compare the effect of packing and non-packing on the healing rate of perianal abscess cavities. Secondary objectives are to assess quality of life, cost effectiveness and rate of abscess recurrence and fistula-in-ano formation. If there is no difference in time to healing and non-packing is shown to be safe, acceptable to the patient and cost effective, this approach may become more widely accepted.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of acute primary perianal abscess
* Have undergone surgical incision and drainage as an emergency

Exclusion Criteria:

* The abscess is the sequelae of concurrent disease or trauma
* Fourniers gangrene is suspected
* Unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Primary Completion 2015-01 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Time to wound healing in days, defined as complete epithelialisation of the abscess cavity. | 1 day to 6 weeks
  time to healing will be assessed in days

SECONDARY OUTCOMES:
Quality of life scores as determined by the Euro QoL EQ-5D-3L | 10 to 14 days
  Quality of life scores as determined by the Euro QoL EQ-5D-3L will be measured at 10-14 days following incision and drainage of abscess

OTHER OUTCOMES:
Abscess recurrence rate | 0 days to 12 months
Fistula-in-ano formation rate | 0 days to 18 months
Cost | 0 days to 18 months